CLINICAL TRIAL: NCT03867136
Title: Refining Multidrug Tuberculosis Treatment with the Ultra Short All Oral Regimen
Brief Title: Refining MDR-TB Treatment (T) Regimens (R) for Ultra(U) Short(S) Therapy(T)
Acronym: TB-TRUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2018-331
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Multidrug Resistant Tuberculosis
Keywords: Multidrug resistant tuberculosis; shorter treatment; all-oral regimen
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PZA sensitivity guided ultra-short all Oral Regimen (Experimental): The PZA sensitivity guided ultra-short regimen consists of two periods of 24-36 weeks. During the first 4-8 weeks(waiting for pyrazinamide drug sensitivity test), the regimen consists of levofloxacin, linezolid, cycloserine, pyrazinamide, and clofazimine. Then based on molecular PZA drug sensitivity results, patients will be in divided into two sub-groups: pyrazinamide-susceptible (PZA-S) patients and pyrazinamide-resistant (PZA-R) patients. The Regimen for PZA-S patients, consisting of levofloxacin, linezolid, cycloserine, and pyrazinamide, are given until the 24th week (prolonged to 28 or 32 weeks if no smear conversion by end of 16th and 20th week). PZA-R sub-group regimen, consisting of levofloxacin, linezolid, cycloserine, and clofazimine given until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week)
  Interventions: Drug: PZA sensitivity guided ultra-short all Oral Regimen
- Standardized Shorter Regimen (Active Comparator): WHO standardized shorter regimen group consists of 36-44 weeks with two phases of treatment. The first is an intensive phase of 16 weeks (extended up a maximum of 20 or 24 weeks in case of lack of smear conversion at the end of 16 or 20 weeks), and included moxifloxacin, amikacin, prothionamide, pyrazinamide, high-dose isoniazid, ethambutol and clofazimine. This is followed by a continuation phase of 20 weeks with the following agents: moxifloxacin, pyrazinamide, ethambutol and clofazimine.
  Interventions: Drug: Standardized Shorter Regimen

INTERVENTIONS:
Drug: PZA sensitivity guided ultra-short all Oral Regimen — Pyrazinamide 1500 mg daily; Levofloxacin ≤50kg 500 mg daily, >50kg 750mg daily; Linezolid: 600 mg daily; Cycloserine ≤50kg 500 mg daily, >50kg 750mg daily; Clofazimine 100 mg daily; All treatment is taken daily;
  Arms: PZA sensitivity guided ultra-short all Oral Regimen
Drug: Standardized Shorter Regimen — Pyrazinamide 1500 mg daily;Levofloxacin 400 mg daily,; Prothionamide ≤50kg 500 mg daily, >50kg 750mg daily; Ethambutol: ≤50kg 750 mg daily, >50kg 1000mg daily; Clofazimine: 100 mg daily; Amikacin 600mg daily; High-dose isoniazid 600mg daily. All treatment is taken daily.
  Arms: Standardized Shorter Regimen

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of a combination of levofloxacin, linezolid, cycloserine and pyrazinamide (or clofazimine if resistant to pyrazinamide) treatments for 24 to 32 weeks (regimen consisted of clofazimine for 36~44 weeks) in subjects with multidrug-resistant tuberculosis (MDR-TB) compared to WHO standardized shorter regimen of 36-44 weeks.

DETAILED DESCRIPTION:
The TB-TRUST is a phaseIII, multicenter, open-label, randomized controlled trial. The purpose of this study is to assess the feasibility of the ultra-short treatment regimen of all-oral anti-TB drugs among selected MDR-TB patients who are susceptible to fluoroquinolones.

A total of 354 participants with MDR-TB will be recruited and followed up until 84 weeks after randomization. During randomization, eligible patients will be assigned to in a 1:1 ratio to one of the following groups: The WHO standardized shorter regimen group and a PZA sensitivity guided ultra-short regimen group.

WHO standardized shorter regimen group consists of 36-44 weeks with two phases of treatment. The first is an intensive phase of 16 weeks (extended up a maximum of 20 or 24 weeks in case of lack of smear conversion at the end of 16 or 20 weeks), and included moxifloxacin, amikacin, prothionamide, pyrazinamide, high-dose isoniazid, ethambutol, and clofazimine. This is followed by a continuation phase of 20 weeks with the following agents: moxifloxacin, pyrazinamide, ethambutol, and clofazimine.

The PZA sensitivity guided ultra-short regimen consists of two periods of 24-36 weeks. During the first 4-8 weeks (waiting for pyrazinamide drug sensitivity test), the regimen consists of levofloxacin, linezolid, cycloserine, pyrazinamide, and clofazimine. Then based on molecular PZA drug sensitivity results, patients will be in divided into two sub-groups: pyrazinamide-susceptible (PZA-S) patients and pyrazinamide-resistant (PZA-R) patients. The Regimen for PZA-S patients, consisting of levofloxacin, linezolid, cycloserine, and pyrazinamide, are given until the 24th week (prolonged to 28 or 32 weeks if no smear conversion by end of 16th and 20th week). PZA-R sub-group regimen, consisting of levofloxacin, linezolid, cycloserine, and clofazimine given until 36th week (prolonged to 40 or 44 weeks if no smear conversion by end of 16th and 20th week)

The primary objective is to compare the treatment success rate without relapse between the WHO standardized shorter regimen group and the PZA sensitivity guided ultra-short regimen group.

The secondary objective is to compare the median time to sputum culture conversion. Safety evaluations performed are the routine lab tests, blood glucose, hearing, vital signs, electrocardiograph (ECG), reporting of adverse events, peripheral neuropathy brief examining with the use of a Brief Peripheral Neuropathy rating scale(BPNS) and ophthalmologic examination, including assessment of visual acuity and color vision，physical examinations and chest CT. Adverse events will be monitored and promptly managed during the whole treatment course.

ELIGIBILITY:
Inclusion Criteria:

1.Willing to participate in trial treatment and follow-up and can give informed consent 2.18-70 years old 3.Has smear-positive pulmonary tuberculosis with initial laboratory results with resistance to rifampicin confirmed by GeneXpert 4.Willing to carry out HIV testing. 5. If you are a non-menopausal woman, agree to use or have used effective contraception during treatment.

6. Have an identifiable address and stay in the area during the study period. 7.Willing to follow the follow-up study procedure after the follow-up.

Exclusion Criteria:

1. Molecular drug resistance test for infected strains resistant to second-line injection;
2. Molecular drug resistance assay for infected strains resistant to fluoroquinolone;
3. Combined extrapulmonary tuberculosis;
4. HIV antibody positive and AIDS patients;
5. Critically ill patients, and according to the judgment of the research physician, it is impossible to survive for more than 16 weeks;
6. Known to be pregnant or breastfeeding;
7. Unable to attend or follow treatment or follow-up time;
8. Can not take oral medications;
9. Patients with impaired liver function (hepatic encephalopathy, ascites; total bilirubin is more than 2 times higher than the upper limit of normal; ALT or AST is more than 5 times the upper limit of normal);
10. Blood muscle spasm is more than 1.5 times the upper limit of normal;
11. The investigator believes that there are any social or medical conditions that expose the subject to a safety hazard;
12. Simultaneously apply the drugs (glucocorticoids, interferons) that affect the efficacy of this study; and apply the following drugs contraindicated with the study drug, including non-steroidal anti-inflammatory drugs, monoamine oxidase inhibitors (phenethyl hydrazine, different Carbofurs et al), direct or indirect sympathomimetic drugs (such as pseudoephedrine), vasopressor drugs (such as adrenaline, norepinephrine), dopamine drugs (such as dopamine, dobutamine), 5 a serotonin reuptake inhibitor, a tricyclic antidepressant, a serotonin 5-HTI receptor antagonist (amitriptyline), meperidine or buspirone.
13. Being allergic or intolerant of any study drug;
14. Currently participating in another drug clinical trial;
15. QTc interval ≥ 500 milliseconds during screening;
16. Hemoglobin is less than 90g/L or platelet is less than 75*10^9/L;
17. Have epilepsy, severe depression, irritability or psychosis；
18. Alchol abuse（drinking more than 64g of ethanol a day for male, 42g for female）.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-08-10 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Treatment success rate of the ultra short regimen | 84 weeks after randomization.
  To compare the treatment success rate without relapse between the PZA sensitivity guided all oral ultra short regimen group and the WHO standardized shorter regimen group. Treatment outcomes will be classified into favourable outcome and unfavourble outcome.

SECONDARY OUTCOMES:
The median time to Sputum Culture Conversion | 12-36 weeks after treatment initiation
  time from treatment initiation to the first of two consecutive negative sputum cultures without an intervening positive culture in liquid media between the ultra short regimen group and the standardized short regimen group;
The frequency of grade 3 or greater adverse events among patients treated with the ultra short regimen | 84 weeks after treatment initiation
  to compare the proportion of patients who experience grade 3 or greater adverse events (graded according to the Division of AIDS severity criteria for adverse events), during treatment or follow-up, on the experimental regimen when compared to the control regimen;

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, PhD, Principal Investigator — Huashan Hospital
Locations (13):
- China (13):
  - The Third People's Hospital of Shenzhen City, Shenzhen, Guangzhou
  - Guiyang Public Health Treatment Center, Guizhou, Guizhou
  - The Sixth People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Chest Hospital, Changsha, Hunan
  - Xuzhou Infectious Disease Hospital, Xuzhou, Jiangsu
  - Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanxi Provincial Tuberculosis Control Institute, Xi’an, Shanxi
  - Southwest Medical University Affiliated Hospital, Luzhou, Sichuan
  - Chest Hospitalof Xinjiang Uygur Autonomous Region of PRC, Ürümqi, Xinjiang
  - Hangzhou Red Cross Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial Center for Disease Control and Prevention, Hangzhou, Zhejiang
  - The Central Hospital of Wenzhou City, Wenzhou, Zhejiang
  - Jiangxi Chest Hospital, Nanchang

REFERENCES:
- [Derived] Weng T, Sun F, Li Y, Chen J, Chen X, Li R, Ge S, Zhao Y, Zhang W. Refining MDR-TB treatment regimens for ultra short therapy (TB-TRUST): study protocol for a randomized controlled trial. BMC Infect Dis. 2021 Feb 17;21(1):183. doi: 10.1186/s12879-021-05870-w. PMID 33596848